CLINICAL TRIAL: NCT01818024
Title: A Three Part, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Repeat Doses of Inhaled and Intravenous GSK2862277 in Healthy Volunteers
Brief Title: A Study to Investigate the Safety Tolerability Pharmacokinetics, and Pharmacodynamics of Inhaled and Intravenous GSK2862277 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 116343
Record Dates: First submitted 2013-02-14; First posted 2013-03-26 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders
Keywords: healthy volunteer; TNFR1; domain antibody; Lung injury
MeSH Terms: conditions — Respiration Disorders; Lung Injury | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part 1: Cohort 1a (Experimental): Single IV dose of GSK2862277 as a continuous infusion over 2 hours.
  Interventions: Drug: Single IV dose of GSK2862277
- Part 1: Cohort 1b (Experimental): Single IV dose of GSK2862277 as a continuous infusion over 3 hours.
  Interventions: Drug: Single IV dose of GSK2862277
- Part 1: Cohort 1c (Experimental): Single IV dose of GSK2862277 as a continuous infusion over 3 hours.
  Interventions: Drug: Single IV dose of GSK2862277
- Part 2: Cohort 2a GSK2862277 (Experimental): Single IV dose of GSK2862277 as a continuous infusion over 1 hour.
  Interventions: Drug: Single IV dose of GSK2862277
- Part 2: Cohort 2a Placebo (Experimental): Matching placebo will be administered as a continuous IV infusion over 1 hour.
  Interventions: Drug: Matching placebo single dose IV infusion
- Part 2: Cohort 2b GSK2862277 (Experimental): Single IH dose of GSK2862277.
  Interventions: Drug: Single IH dose of GSK2862277
- Part 2: Cohort 2b Placebo (Experimental): Matching placebo will be administered.
  Interventions: Drug: Matching placebo single dose IH
- Part 3: Cohort 3a GSK2862277 (Experimental): IV dose of GSK2862277 (decided from Part 2) as a continuous infusion over 1 hour for daily 5 days.
  Interventions: Drug: Repeat IV dose of GSK2862277
- Part 3: Cohort 3a Placebo (Experimental): Matching placebo will be administered as IV infusion over 1 hour daily for 5 days.
  Interventions: Drug: Matching placebo repeat dose IV infusion
- Part 3: Cohort 3b GSK2862277 (Experimental): Repeat IH dose of GSK2862277 (decided from Part 2) daily for 5 days.
  Interventions: Drug: Repeat IH dose selected of GSK2862277 from Part 2
- Part 3: Cohort 3b Placebo (Experimental): Matching placebo will be administered as IH daily for 5 days.
  Interventions: Drug: Matching placebo repeat dose IH

INTERVENTIONS:
Drug: Single IV dose of GSK2862277 — GSK2862277 solution available in a 40 mg vial for IV administration.
  Arms: Part 1: Cohort 1a; Part 1: Cohort 1b; Part 1: Cohort 1c; Part 2: Cohort 2a GSK2862277
Drug: Matching placebo single dose IV infusion — Matching placebo solution available for IV administration.
  Arms: Part 2: Cohort 2a Placebo
Drug: Single IH dose of GSK2862277 — GSK2862277 nebulised solution available in a 40 mg vial for IH administration.
  Arms: Part 2: Cohort 2b GSK2862277
Drug: Matching placebo single dose IH — Matching placebo nebulised solution available for IH administration.
  Arms: Part 2: Cohort 2b Placebo
Drug: Repeat IV dose of GSK2862277 — GSK2862277 solution available in a 40 mg vial for IV administration.
  Arms: Part 3: Cohort 3a GSK2862277
Drug: Matching placebo repeat dose IV infusion — Matching placebo solution available for IV administration.
  Arms: Part 3: Cohort 3a Placebo
Drug: Repeat IH dose selected of GSK2862277 from Part 2 — GSK2862277 nebulised solution available in a 40 mg vial for IH administration.
  Arms: Part 3: Cohort 3b GSK2862277
Drug: Matching placebo repeat dose IH — Matching placebo nebulised solution available for IH administration.
  Arms: Part 3: Cohort 3b Placebo

SUMMARY:
This will be a 3 part study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and repeat doses of GSK2862277 administered via inhalation (IH) or intravenous (IV) routes in healthy subjects.

Part 1 of this study will involve an initial assessment of safety, tolerability and pharmacokinetics of GSK286227, via single escalating intravenous doses, compared to a predecessor molecule, GSK1995057. After completion of Part 1 an interim data review will occur which will assess key comparability criteria to inform progression to Part 2 of the study.

Part 2 of the study will involve single doses of GSK2862277 at a level predicted to be at or close to therapeutic dose levels. Part 2 will investigate both intravenous and inhaled routes of administration, in sequential manner, respectively. An interim data review will also occur after completion of Part 2, where all data accumulated previously will be assessed to examine appropriateness to progress to Part 3.

Part 3 of the study will involve 5 days of repeat dosing via both inhaled and intravenous routes using the same dose administered in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subject is positive at screening for HAVH autoantibodies against GSK1995057 (Part 1 only).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2013-10-25 (Actual); Study Completion 2013-10-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single IV or IH dose of GSK2862277 assessed by number of subjects with adverse events (AE)s in Part 1 and Part 2 | Up to 42 days
  Safety and tolerability parameters will include recording of adverse events (AEs), throughout the study.
Safety and tolerability of repeat IV or IH dose of GSK2862277 assessed by number of subjects with AEs in Part 3 | Up to 42 days
  Safety and tolerability parameters will include recording of AEs, throughout the study.
Safety and tolerability of single IV or IH dose of GSK2862277 assessed by laboratory tests in Part 1 and Part 2 | Up to 42 days
  Laboratory tests will include haemogram, clinical chemistry, urine examination.
Safety and tolerability of repeat IV or IH dose of GSK2862277 as assessed by laboratory tests in Part 3 | Up to 42 days
  Laboratory tests will include haemogram, clinical chemistry, urine examination.
Safety and tolerability of single IV or IH dose of GSK2862277 assessed by vital signs in Part 1 and Part 2 | Up to 42 days
  Vital signs will include blood pressure (BP), heart rate respiration rate and body temperature.
Safety and tolerability of repeat IV or IH dose of GSK2862277 assessed by vital signs in Part 3 | Up to 42 days
  Vital signs will include BP, heart rate respiration rate and body temperature.
Safety and tolerability of single IV or IH dose of GSK2862277 assessed by ECG in Part 1 and Part 2 | Up to 42 days
  Safety data will include electrocardiogram (ECG) readings obtained at each timepoint during the study.
Safety and tolerability of repeat IV or IH dose of GSK2862277 assessed by ECG in Part 3 | Up to 42 days
  Safety data will include ECG readings obtained at each timepoint during the study.
Safety and tolerability of single IV or IH dose of GSK2862277 assessed by spirometry monitoring in Part 1 and Part 2 | Up to 42 days
  Spirometry monitoring will include forced expiratory volume in one second (FEV1) and forced vital capacity (FVC).
Safety and tolerability of repeat IV or IH dose of GSK2862277 assessed by spirometry monitoring in Part 3 | Up to 42 days
  Spirometry monitoring will include FEV1 and FVC.
Safety and tolerability of single IV dose of GSK2862277 as assessed by measurement of plasma cytokines in Part 1 | Up to 42 days
  Blood samples will be collected for assessment of plasma cytokines.
Immunogenicity in subjects receiving single IV or IH dose of GSK2862277 in Part 1 and Part 2 | Up to 60 days
  Presence of anti GSK2862277 binding antibodies will be evaluated.
Immunogenicity in subjects receiving repeat IV or IH dose of GSK2862277 in Part 3 | Up to 60 days
  Presence of anti GSK2862277 binding antibodies will be evaluated.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters in subjects receiving single IV or IH dose of GSK2862277 in Part 1 and Part 2 | Up to 48 hours post dose
  The blood samples will be collected for plasma concentrations of GSK2862277.
PK parameters in subjects receiving repeat IV dose of GSK2862277 in Part 3 Cohort 3a | Up to 48 hours post last dose
  The blood samples will be collected for plasma concentrations of GSK2862277.
PK parameters in subjects receiving repeat IH dose of GSK2862277 in Part 3 Cohort 3b | Up to 48 hours post last dose
  The blood samples will be collected for plasma concentrations of GSK2862277
PK parameters in subjects receiving single IV dose of GSK2862277 in Part 1 | Up to 48 hours post last dose
  The PK parameters will be compared with historic GSK1995057 PK data in Part 1
Pharmacodynamic and immune function biomarkers in serum of subjects receiving single IV or IH dose of GSK2862277 in Part 1 and Part 2 | Up to 48 hours post last dose
  The pharmacodynamic and immune function biomarkers in serum.
Pharmacodynamic and immune function biomarkers in serum of subjects receiving repeat IV or IH dose of GSK2862277in Part 3 | Up to 48 hours post last dose
  The pharmacodynamic and immune function biomarkers in serum.
Change from baseline in IL-8 expression in ex vivo WBA in subjects receiving single IV 0.05 mg/kg dose of GSK2862277 in Part 1 in Cohort1c | Up to 12 hours post dose
  IL-8 expression in ex vivo whole blood essay (WBA).
Composite of urine parameters in subjects receiving single IV 2 mg/kg dose of GSK2862277 in Part 2 in Cohort 2a | Up to 48 hours post dose
  The urine samples will be collected for urine concentrations of GSK2862277.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Cordy JC, Morley PJ, Wright TJ, Birchler MA, Lewis AP, Emmins R, Chen YZ, Powley WM, Bareille PJ, Wilson R, Tonkyn J, Bayliffe AI, Lazaar AL. Specificity of human anti-variable heavy (VH ) chain autoantibodies and impact on the design and clinical testing of a VH domain antibody antagonist of tumour necrosis factor-alpha receptor 1. Clin Exp Immunol. 2015 Nov;182(2):139-48. doi: 10.1111/cei.12680. Epub 2015 Sep 11. PMID 26178412
- See also: Results for study 116343 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116343?search=study&search_terms=116343#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116343 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register